CLINICAL TRIAL: NCT00721110
Title: Effects of Perioperative Lidocaine and Ketamine Infusions on Acute Functional Recovery After Abdominal Hysterectomy
Brief Title: Lidocaine and Ketamine in Abdominal Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Futility
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08-454
Record Dates: First submitted 2008-07-21; First posted 2008-07-23 (Estimated); Results first posted 2017-07-26 (Actual); Last update posted 2017-07-26 (Actual); Status verified 2017-04

CONDITIONS: Abdominal Hysterectomy (& Wertheim)
Keywords: pain control; nausea; surgery recovery
MeSH Terms: conditions — Agnosia; Nausea | interventions — Lidocaine; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Lidocaine (Active Comparator): Intravenous Lidocaine Group - Lidocaine is administered intravenously throughout surgery and during the 24 hours following surgery
  Interventions: Drug: Lidocaine
- Placebo (Placebo Comparator): A lidocaine placebo is administered intravenously throughout surgery and during the 24 hours after surgery.
  Interventions: Drug: Placebo
- Ketamine (Active Comparator): Intravenous Ketamine Group - Ketamine is administered intravenously throughout surgery and during the 24 hours following surgery
  Interventions: Drug: Ketamine
- ketamine + Lidocaine (Active Comparator): both ketamine and Lidocaine are administered intravenously throughout surgery and during the 24 hours after surgery.
  Interventions: Drug: Ketamine + Lidocaine

INTERVENTIONS:
Drug: Lidocaine — Upon general anesthesia induction, lidocaine (1.5 mg/kg) will be given. Lidocaine infusion of 2 mg/kg/hour, to a maximum of 200 mg/hour during The lidocaine infusion will be reduced to 1.3 mg/kg/hour, to a maximum of 133 mg/hour, at skin closure and discontinued 24 hours postoperatively.
  Arms: Lidocaine
Drug: Placebo — Placebo boluses and infusions will be substituted
  Arms: Placebo
Drug: Ketamine — Ketamine (0.25 mg/kg) will be given followed by an infusion of ketamine (0.25 mg/kg/hour) up to 25 mg/hour. The ketamine infusion will be reduced to 0.12 mg/kg/hour up to a maximum of 12 mg/hour at skin closure and discontinued 24 hours postoperatively.
  Arms: Ketamine
Drug: Ketamine + Lidocaine — both Ketamine and Lidocaine will be given
  Arms: ketamine + Lidocaine

SUMMARY:
This study is being done to determine if combined infusions of lidocaine and ketamine is better than a lidocaine or ketamine infusion alone, or to placebo in improving recovery after abdominal hysterectomy. Participants will be randomized into one of four groups. Evaluations will be done through walking tests, pain and fatigue questionnaires and blood tests.

DETAILED DESCRIPTION:
Subjects undergoing abdominal hysterectomy surgery are randomized into one of four groups: Intravenous Lidocaine, Intravenous Ketamine, Intravenous Lidocaine and Ketamine or Placebo. Subjects will perform a six-minute walk test prior to surgery and on the second day postoperatively. After surgery and on days 1 and 2 after surgery, subjects will rate their pain. On day 1 postoperatively, subjects will rate their fatigue. On postoperative days 1 and 2 incisional pain will be analysed using von Frey filaments. Two hours after surgery, 10 ml of venous blood will be sampled for cytokine analysis. Telephone follow up will take place 6 and 12 months postoperatively to access pain and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years old and less than 75 years years old
* Horizontal abdominal incision

Exclusion Criteria:

* Emergency or urgent procedure
* Preexisting chronic pain (at any site) requiring treatment
* Contraindication to any study medication (ketamine or lidocaine)
* History of significant Axis I psychiatric disease (major depressive disorder, bipolar disorder, schizophrenia, etc.)
* Significant hepatic (ALT or AST > 2 times normal) or renal (serum creatinine > 2 mg/dl) impairment
* Seizure disorder requiring medication within past 2 years
* Planned spinal or epidural anesthesia or analgesia

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-07; Primary Completion 2010-10 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Grady, MD, Principal Investigator — The Cleveland Clinic; Daniel I Sessler, MD, Study Chair — The Cleveland Clinic
Locations (1):
- Cleveland Clinic/Hillcrest Hospital, Mayfield Heights, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a factorial study design with 64 patients randomized to 2 treatments each: lidocaine or placebo and ketamine or placebo. Each treatment was analyzed separately (i.e., lidocaine versus placebo and ketamine versus placebo separately). Though there are 4 distinct groups, the same 64 patients are in both lidocaine and ketamine analyses.
Groups:
- Lidocaine/Ketamine: Intravenous Lidocaine + Ketamine Group
  Lidocaine was given as a bolus (1.5 mg/kg), followed by an infusion of 2 mg/kg/h for the first 2 hours, and then 1.2 mg/kg/h for 24 postoperative hours.
  Ketamine was given as a bolus (0.35 mg/kg), followed by ketamine infusion of 0.2 mg/kg/h for the first 2 hours, and then 0.12 mg/kg/h for 24 postoperative hours.
  Medication doses were based on actual patient body weight to a maximum of 150% of ideal body weight based on the formula: 49 kg + 0.6 kg for each centimeter of height exceeding 152 centimeters
- Lidocaine: Intravenous lidocaine Group - Lidocaine was given as a bolus (1.5 mg/kg), followed by an infusion of 2 mg/kg/h for the first 2 hours, and then 1.2 mg/kg/h for 24 postoperative hours.
- Ketamine: Intravenous Ketamine Group - Ketamine is administered intravenously throughout surgery and during the 24 hours following surgery
  Ketamine: Upon induction of anesthesia, a bolus of ketamine (0.25mg/kg) will be given followed by an infusion of ketamine (0.25mg/kg/hour) up to 25 mg/hour. The ketamine infusion will be reduced to 0.12 mg/kg/hour up to a maximum of 12 mg/hour at skin closure and discontinued 24 hours postoperatively.
- Placebo: A placebo is administered intravenously throughout surgery and during the 24 hours after surgery.
  A placebo infusion will be substituted for the ketamine or lidocaine not given
Period: Overall Study
Arm/Group | Lidocaine/Ketamine | Lidocaine | Ketamine | Placebo
Started | 16 | 16 | 16 | 16
Completed | 15 | 16 | 15 | 16
Not Completed | 1 | 0 | 1 | 0
Not completed — Ultram use | 1 | 0 | 0 | 0
Not completed — vertical incision | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Lidocaine/Ketamine: Intravenous Lidocaine and Ketamine Group -
  Lidocaine was given as a bolus (1.5 mg/kg), followed by an infusion of 2 mg/kg/h for the first 2 hours, and then 1.2 mg/kg/h for 24 postoperative hours. Ketamine was given as a bolus (0.35 mg/kg), followed by ketamine infusion of 0.2 mg/kg/h for the first 2 hours, and then 0.12 mg/kg/h for 24 postoperative hours. Medication doses were based on actual patient body weight to a maximum of 150% of ideal body weight based on the formula: 49 kg + 0.6 kg for each centimeter of height exceeding 152 centimeters.
- Lidocaine: Intravenous lidocaine Group - A lidocaine is administered intravenously through out surgery and 24 hours after surgery.
  Lidocaine was given as a bolus (1.5 mg/kg), followed by an infusion of 2 mg/kg/h for the first 2 hours, and then 1.2 mg/kg/h for 24 postoperative hours.
- Total: Total of all reporting groups
Arm/Group | Lidocaine/Ketamine | Lidocaine | Ketamine | Placebo | Total
Number analyzed (Participants) | 15 | 16 | 15 | 16 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (7) | 46 (7) | 46 (9) | 47 (8) | 46 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 15 | 16 | 62
  Male | 0 | 0 | 0 | 0 | 0
American Society of Anesthesiologists Physical Status [Number; unit: participants] — American Society of Anesthesiologists Physical Status applied to each patient ranging from I to VI. The scale is defined as follows:
  I: A normal healthy patient II: A patient with mild systemic disease III: A patient with severe systemic disease IV: A patient with severe systemic disease that is a constant threat to life V: A moribund patient who is not expected to survive without the operation VI: A declared brain-dead patient whose organs are being removed for donor purposes
  participants
    A normal healthy patient | 0 | 0 | 2 | 0 | 2
    A patient with mild systemic disease | 14 | 13 | 10 | 15 | 52
    A patient with severe systemic disease | 1 | 3 | 3 | 1 | 8
Body Mass Index [Mean (Standard Deviation); unit: kg per meters squared] | 28 (6) | 29 (6) | 29 (10) | 28 (6) | 29 (7)
Preoperative 6-MWD [Mean (Standard Deviation); unit: m] | 318 (47) | 320 (44) | 304 (41) | 338 (52) | 320 (47)

OUTCOME MEASURES:

1. Primary Outcome: The Effects of Lidocaine and Ketamine on Functional Recovery Assessed by 6 Minute Walk Test on Postoperative Day Two
Description: The effects of lidocaine and ketamine on functional recovery assessed by 6 minute walk test on postoperative day two after hysterectomy. This outcome measures return to ambulation after surgery.
Time Frame: postoperative day 2
Measure: Mean (Standard Deviation); unit: meters
Groups:
- Nonlidocaine: Intravenous Nonlidocaine Group - A lidocaine placebo is administered intravenously through out surgery and 24 hours after surgery.
  Placebo boluses and infusions will be substituted for the lidocaine
- Nonketamine: A ketamine placebo is administered intravenously throughout surgery and during the 24 hours after surgery.
  A placebo infusion will be substituted for the ketamine not given
Arm/Group | Lidocaine | Nonlidocaine | Ketamine | Nonketamine
Number analyzed (Participants) | 31 | 31 | 30 | 32
meters | 202 (66) | 202 (73) | 193 (77) | 210 (61)
Statistical Analysis 1: Comparison: Lidocaine vs Nonlidocaine; The effect of lidocaine on 6-minute walk distance on the 2nd postoperative morning was assessed using analysis of covariance. We expected the control group's mean 6-minute walk distance to be 300 meters with a standard deviation (SD) of about 20% of the mean for each group. Assuming a correlation of 0.5 between baseline and 2nd postoperative day, a maximum 128 total patients (32 for each group) was needed to have 80% power at the 0.025 significance level to detect effects of 36 meters or more; Test type: Superiority or Other; p = 0.96, ANCOVA — Significant if P < 0.003 for efficacy and P > 0.5311 for futility; 97.5% confidence intervals adjusted for group sequential design to maintain the overall alpha of 0.025 for each primary intervention; Adjusted for baseline 6-minute walk distance; Mean Difference (Final Values) = 0.93, 97.5% CI 2-sided [-52 to 54]
Statistical Analysis 2: Comparison: Ketamine vs Nonketamine; The effect of ketamine on 6-minute walk distance on the 2nd postoperative morning was assessed using analysis of covariance. We expected the control group's mean 6-minute walk distance to be 300 meters with a standard deviation (SD) of about 20% of the mean for each group. Assuming a correlation of 0.5 between baseline and 2nd postoperative day, a maximum 128 total patients (32 for each group) was needed to have 80% power at the 0.025 significance level to detect effects of 36 meters or more; Test type: Superiority or Other; p = 0.54, ANCOVA — 97.5% confidence interval adjusted for group sequential design (using confidence coefficient of 2.97) to maintain theoverall α of 0.025 for each primary intervention and 0.05 for the trial; Adjusted for baseline 6-minute walk distance; Mean Difference (Final Values) = -11, 97.5% CI 2-sided [-65 to 44]

2. Secondary Outcome: Verbal Response Pain Scores (VRS) at PACU Admission and Discharge as Well as Mornings and Afternoons of Postoperative Days 1 and 2
Description: Verbal response pain scores (VRS) at PACU admission and discharge as well as mornings and afternoons of postoperative days 1 and 2. VRS scale ranges from 0 to 10, with 0 denoting no pain and 10 denoting worst possible pain.
Time Frame: PACU admission and discharge, postoperative mornings and afternoons on days 1 and 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lidocaine | Nonlidocaine | Ketamine | Nonketamine
Number analyzed (Participants) | 31 | 31 | 30 | 32
units on a scale
  PACU admit | 6.2 (3.3) | 7.1 (2.5) | 6.4 (3.4) | 6.9 (2.5)
  PACU discharge | 4.0 (2.3) | 4.9 (1.9) | 4.6 (2.4) | 4.3 (1.9)
  POD 1 | 4.0 (1.8) | 3.3 (2.2) | 3.7 (2.2) | 3.6 (1.7)
  POD 2 | 3.1 (1.7) | 2.9 (1.9) | 3.1 (2.1) | 2.8 (1.4)
Statistical Analysis 1: Comparison: Lidocaine vs Nonlidocaine; Groups compared on VRS scores at PACU admit using a t test; Test type: Superiority or Other; p = 0.20, t-test, 2 sided — 97.5% confidence intervals (CIs) adjusted for group sequential design (using confidence coefficient of 2.97) to maintain the overall α of 0.025 for each intervention and 0.05 for the trial; Mean Difference (Final Values) = -1.0, 97.5% CI 2-sided [-3.3 to 1.3]
Statistical Analysis 2: Comparison: Ketamine vs Nonketamine; Ketamine compared to placebo at PACU admit using a t test; Test type: Superiority or Other; p = 0.54, t-test, 2 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.5, 97.5% CI 2-sided [-2.8 to 1.9]
Statistical Analysis 3: Comparison: Lidocaine vs Nonlidocaine; Lidocaine versus nonlidocaine on pain severity at postoperative care unit discharge was assessed using a t test; Test type: Superiority or Other; p = 0.11, t-test, 2 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.9, 97.5% CI 2-sided [-2.5 to 0.8]
Statistical Analysis 4: Comparison: Ketamine vs Nonketamine; Ketamine versus nonketamine on postoperative care unit discharge pain severity was assessed using a t test; Test type: Superiority or Other; p = 0.56, t-test, 2 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.3, 97.5% CI 2-sided [-1.4 to 2.0]
Statistical Analysis 5: Comparison: Lidocaine vs Nonlidocaine; Lidocaine versus nonlidocaine on postoperative day 1 pain severity assessed using a t test; Test type: Superiority or Other; p = 0.20, t-test, 2 sided — [p-value comment as in outcome 2, analysis 1]; Median Difference (Final Values) = 0.6, 97.5% CI 2-sided [-0.9 to 2.2]
Statistical Analysis 6: Comparison: Ketamine vs Nonketamine; Ketamine versus nonketamine on postoperative day 1 pain severity was assessed using a t test; Test type: Superiority or Other; p = 0.79, t-test, 2 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.1, 97.5% CI 2-sided [-1.4 to 1.7]
Statistical Analysis 7: Comparison: Lidocaine vs Nonlidocaine; Lidocaine versus nonlidocaine on postoperative day 2 pain severity was assessed using a t test; Test type: Superiority or Other; p = 0.55, t-test, 2 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.3, 97.5% CI 2-sided [-1.1 to 1.7]
Statistical Analysis 8: Comparison: Ketamine vs Nonketamine; Ketamine versus nonketamine on postoperative day 2 pain severity was assessed using a t test; Test type: Superiority or Other; p = 0.47, t-test, 2 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.3, 97.5% CI 2-sided [-1.1 to 1.8]

3. Secondary Outcome: Total Opioid Consumption at PACU Admission and Discharge as Well as Mornings of Postoperative Days 1 and 2
Time Frame: intraoperative through postoperative day 2
Measure: Median (Inter-Quartile Range); unit: milligram morphine sulfate equivalents
Arm/Group | Lidocaine | Nonlidocaine | Ketamine | Nonketamine
Number analyzed (Participants) | 31 | 31 | 30 | 32
milligram morphine sulfate equivalents
  intraoperative | 20 [15 to 30] | 20 [19 to 30] | 20 [15 to 26] | 23 [20 to 30]
  postoperative care unit | 20 [7 to 27] | 23 [18 to 27] | 20 [7 to 27] | 23 [19 to 27]
  postoperative day 1 | 23 [15 to 48] | 22 [13 to 50] | 21 [12 to 48] | 23 [17 to 47]
  postoperative day 2 | 10 [3 to 18] | 6 [2 to 15] | 9 [3 to 20] | 8 [3 to 14]
Statistical Analysis 1: Comparison: Lidocaine vs Nonlidocaine; Lidocaine versus nonlidocaine on intraoperative opioid consumption was assessed using the Wilcoxon rank sum test; Test type: Superiority or Other; p = 0.63, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 2, analysis 1]; Median Difference (Final Values) = 0, 97.5% CI 2-sided [-7 to 7]
Statistical Analysis 2: Comparison: Ketamine vs Nonketamine; Ketamine versus nonketamine on intraoperative opioid consumption was assessed using a Wilcoxon rank sum test; Test type: Superiority or Other; p = 0.27, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 2, analysis 1]; Median Difference (Final Values) = -2, 97.5% CI 2-sided [-10 to 5]
Statistical Analysis 3: Comparison: Lidocaine vs Nonlidocaine; Lidocaine versus nonlidocaine on postoperative care unit opioid consumption was assessed using a Wilcoxon rank sum test; Test type: Superiority or Other; p = 0.28, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 2, analysis 1]; Median Difference (Final Values) = -3, 97.5% CI 2-sided [-15 to 5]
Statistical Analysis 4: Comparison: Ketamine vs Nonketamine; Ketamine versus nonketamine on postoperative care unit opioid consumption was assessed using a Wilcoxon rank sum test; Test type: Superiority or Other; p = 0.22, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 2, analysis 1]; Median Difference (Final Values) = -4, 97.5% CI 2-sided [-15 to 4]
Statistical Analysis 5: Comparison: Lidocaine vs Nonlidocaine; Lidocaine versus nonlidocaine on postoperative day 1 opioid consumption was assessed using a Wilcoxon rank sum test; Test type: Superiority or Other; p = 0.76, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 2, analysis 1]; Median Difference (Final Values) = 2.5, 97.5% CI 2-sided [-13 to 21]
Statistical Analysis 6: Comparison: Ketamine vs Nonketamine; Ketamine versus nonketamine on postoperative day 1 opioid consumption was assessed using a Wilcoxon rank sum test; Test type: Superiority or Other; p = 0.66, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 2, analysis 1]; Median Difference (Final Values) = -3, 97.5% CI 2-sided [-19 to 14]
Statistical Analysis 7: Comparison: Lidocaine vs Nonlidocaine; Lidocaine versus nonlidocaine on postoperative day 2 opioid consumption was assessed using a Wilcoxon rank sum test; Test type: Superiority or Other; p = 0.30, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 2, analysis 1]; Median Difference (Final Values) = 2.5, 97.5% CI 2-sided [-5 to 10]
Statistical Analysis 8: Comparison: Ketamine vs Nonketamine; Ketamine versus nonketamine on postoperative day 2 opioid consumption was assessed using a Wilcoxon rank sum test; Test type: Superiority or Other; p = 0.79, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 2, analysis 1]; Median Difference (Final Values) = 0, 97.5% CI 2-sided [-5 to 8]

4. Secondary Outcome: Presence of Nausea and Vomiting After Two Hours in the PACU and the First Postoperative Day
Time Frame: 2 hours after surgery, on postoperative day 1
Measure: Number; unit: percentage of participants
Arm/Group | Lidocaine | Nonlidocaine | Ketamine | Nonketamine
Number analyzed (Participants) | 31 | 31 | 30 | 32
percentage of participants
  Nausea, PACU | 32 | 26 | 30 | 28
  Nausea, POD 1 | 55 | 48 | 53 | 50
  Vomiting, PACU | 6 | 19 | 10 | 16
  Vomiting, POD 1 | 23 | 16 | 23 | 16
Statistical Analysis 1: Comparison: Lidocaine vs Nonlidocaine; Lidocaine versus nonlidocaine on PACU (postoperative care unit) nausea assessed using Pearson chi square test; Test type: Superiority or Other; p = 0.58, Chi-squared — [p-value comment as in outcome 2, analysis 1]; Risk Ratio (RR) = 0.06, 97.5% CI 2-sided [-0.28 to 0.41] — numerator: lidocaine; denominator: control
Statistical Analysis 2: Comparison: Ketamine vs Nonketamine; Ketamine versus nonketamine on PACU (postoperative care unit) nausea assessed using Pearson chi square test; Test type: Superiority or Other; p = 0.87, Chi-squared — [p-value comment as in outcome 2, analysis 1]; Risk Ratio (RR) = 0.02, 97.5% CI 2-sided [-0.32 to 0.36] — Numinator: ketamine; denominator: nonketamine
Statistical Analysis 3: Comparison: Lidocaine vs Nonlidocaine; Lidocaine versus nonlidocaine on POD 1 (first postoperative day) nausea assessed using Pearson chi square test; Test type: Superiority or Other; p = 0.61, Chi-squared — [p-value comment as in outcome 2, analysis 1]; Risk Ratio (RR) = 0.06, 97.5% CI 2-sided [-0.31 to 0.44]
Statistical Analysis 4: Comparison: Ketamine vs Nonketamine; Ketamine versus nonketamine on POD 1(first postoperative day) nausea assessed using Pearson chi square test; Test type: Superiority or Other; p = 0.79, Chi-squared — [p-value comment as in outcome 2, analysis 1]; Risk Ratio (RR) = 0.03, 97.5% CI 2-sided [-0.34 to 0.41]
Statistical Analysis 5: Comparison: Lidocaine vs Nonlidocaine; Lidocaine versus nonlidocaine on PACU (postoperative care unit) vomiting assessed using Pearson chi square test; Test type: Superiority or Other; p = 0.26, Chi-squared — [p-value comment as in outcome 2, analysis 1]; Risk Ratio (RR) = -0.13, 97.5% CI 2-sided [-0.38 to 0.12]
Statistical Analysis 6: Comparison: Ketamine vs Nonketamine; Ketamine versus nonketamine on PACU (postoperative care unit) vomiting assessed using a Pearson chi square test; Test type: Superiority or Other; p = 0.71, Chi-squared — [p-value comment as in outcome 2, analysis 1]; Risk Ratio (RR) = -0.06, 97.5% CI 2-sided [-0.31 to 0.19]
Statistical Analysis 7: Comparison: Lidocaine vs Nonlidocaine; Lidocaine versus nonlidocaine on postoperative day 1 vomiting assessed using a Pearson chi square test; Test type: Superiority or Other; p = 0.52, Chi-squared — [p-value comment as in outcome 2, analysis 1]; Risk Ratio (RR) = 0.06, 97.5% CI 2-sided [-0.23 to 0.36]
Statistical Analysis 8: Comparison: Ketamine vs Nonketamine; Ketamine versus nonketamine on postoperative day 1 vomiting assessed using Pearson chi square test; Test type: Superiority or Other; p = 0.44, Chi-squared; Risk Ratio (RR) = 0.07, 97.5% CI 2-sided [-0.22 to 0.38]

5. Secondary Outcome: Verbal Response Fatigue Score on Postoperative Day 1
Description: Verbal response fatigue score on postoperative day 1. Verbal response fatigue score measured on a scale ranging from 0 to 10, where 0 is no fatigue and 10 is the worst possible fatigue.
Time Frame: postoperative day 1
Population: 11 patients had missing POD 1 fatigue scores (e.g., 11 for lidocaine vs. nonlidocaine and 11 for ketamine vs. nonketamine).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lidocaine | Nonlidocaine | Ketamine | Nonketamine
Number analyzed (Participants) | 26 | 25 | 24 | 27
units on a scale | 7.2 (2.5) | 7.2 (2.4) | 7.4 (2.6) | 7.0 (2.3)
Statistical Analysis 1: Comparison: Lidocaine vs Nonlidocaine; Lidocaine was compared to nonlidocaine on mean VRS fatigue score using a t test; Test type: Superiority or Other; p = 0.96, t-test, 2 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.03, 97.5% CI 2-sided [-2.14 to 2.2]
Statistical Analysis 2: Comparison: Ketamine vs Nonketamine; Ketamine was compared to nonketamine on mean VRS fatigue score using a t test; Test type: Superiority or Other; p = 0.59, t-test, 2 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.3, 97.5% CI 2-sided [-1.80 to 2.57]

ADVERSE EVENTS:
Groups:
- Placebo: placebo is administered intravenously through out surgery and 24 hours after surgery.
- Ketamine + Lidocaine: both ketamine and Lidocaine administered intravenously throughout surgery and during the 24 hours after surgery.
Arm/Group | Lidocaine | Placebo | Ketamine | Ketamine + Lidocaine
All-Cause Mortality (participants affected / at risk) | 16/16 | 16/16 | 15/15 | 15/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes